CLINICAL TRIAL: NCT01682252
Title: Cellular Analysis of Blood Suctioned During Surgery for Musculoskeletal Tumors
Brief Title: Analysis of Blood During Surgery for Musculoskeletal Tumors
Status: Terminated | Type: Observational
Why Stopped: investigators felt sufficient data has been collected
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Anesthesia, Yuriy Gubenko, MD Assistant Professor, Rutgers, The State University of New Jersey
Other Study IDs: 01201000247
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Musculoskeletal Tumors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- musculoskeletal tumors: all patients undergoing surgery for musculoskeletal tumors

SUMMARY:
This study is being done as the doctor investigators would like to lessen the amount of blood transfusions given to patients. Patients who receive blood transfusions have a greater chance of developing complications after surgery. There is a device called the Cell Saver that allows the doctors to process blood that is lost during surgery and return it to the patient. This lessens the amount of transfused blood the patients receive. This device is not used for patients undergoing surgery for muscular skeletal tumors.The investigators are not sure whether tumor cells are present in the blood which is lost during the course of an operation like yours. The goal of this study is to see if we lessen the amount of blood transfusions given to patients who may have tumor or cancerous cells present in their blood. One way to do this is to test the blood that is circulating in your veins and also to test the blood which is lost during the course of your operation

DETAILED DESCRIPTION:
Allogenic Blood transfusions are associated with numerous complications from simple uticaria to serious transmissible diseases. While improved testing has significantly decreased the incidence of AIDS and hepatitis C to approximately 1:2,000,000 units tested; hepatitis B approximately 1:200,000 units tested, more frequent complications occur secondary to immunomodulation, which results in making infections more common. These are not due to infected blood, but develop because of changes in patients' immune system after having received an allogenic red blood cell transfusion. The relative risk for developing an infection is 1.6 for 1-3 red blood cell units and 3.6 for patients who receive more than 3 red cell units. Patients who receive transfusions have a 52% greater risk of developing pneumonia and a 35% greater risk of developing a urinary tract infection. On average, hospitalization costs $14,000 more for patients with a serious infection. These infections prolong the length of hospitalization after surgery and may even result in death.2 Other complications of transfusion include Transfusion Related Acute Lung Injury which causes at least 5300 TRALI reactions per year in the US alone, and approximately 500 deaths. In fact, just one donor whose blood triggered a TRALI death was found on review of records to have caused 14 previous cases of TRALI. Other serious complications include Adult Respiratory Distress Syndrome, and transfusion reactions. As a group, these complications of transfusion result in increased morbidity and mortality. Therefore, it is in the best interest of patients to decrease the amount of allogenic blood transfused (from other individuals). To prevent this, surgeons employ the use of a Cell Saver (CS) during surgery which collects the patient's own blood from the operative field and washes it. This blood is then re-infused into the patient's intravenous, minimizing the need for transfusion of blood from the blood bank.

Despite the benefits of the cell saver, it is not used in patients who have malignancy due to concern that the tumor cells may spread systemically via the blood. Due to the nature of musculoskeletal tumor resections there is often significant blood loss. Dissection is regularly through the muscles rather than around muscular intervals, which can result in significant bleeding. The goal of this study is to determine the presence or absence of tumor cells in the blood suctioned from the surgical field. Pending the outcome, consideration will be made to go forward with a second study to determine if cell saver could be used in patients with malignancy undergoing surgery.

It is unclear whether tumor cells are present in the blood suctioned from an extremity malignancy resection. It is also unknown if the processing of blood suctioned would remove tumor cells from the blood to be transfused. If no tumor cells are found in the blood after processing then transfusion of this blood would likely be safe. This could result in decreased blood transfusions in this patient population. This would not only decrease risk to these patients, it would also improve the blood supply, ensuring that blood is available for other patients who require it. This work is highly significant as it would both improve safety in this patient population and improve the blood supply. Data collected will include the patient's diagnosis, the presence or absence of metastatic disease, whether they have been previously treated with chemotherapy or radiation and the dates of that treatment. Patients will undergo surgery and anesthesia in the usual manner. Three sets of specimens approximately 4mL each would be taken; one from a peripheral line prior to opening the skin, the second sample will be taken from the surgical field or suction canister during the tumor resection the third from the surgical field or suction canister shortly before the tumor is removed. These samples will be taken to Dr. Fitzhugh's laboratory for slide staining.

Patients who are determined by their surgeon and/or anesthesiologist to require blood will be administered blood processed by the University Hospital Blood Bank using standard transfusion protocols. No blood taken from the patient or the operative field will be transfused.

There are no significant risks in this study. Roughly 2 ml of blood is required for the total number of slides (2-4) that would be prepared per tube. This amount of blood 12 mL is less than one tablespoon and does not pose significant risk to the patient nor does it increase the likelihood of transfusion. Slides will be stained using the Diff-Quik staining method, a method similar to the Wright-Giemsa staining used in hematology laboratories. The technique is rapid (requires only 3 minutes per submitted sample) and inexpensive. Slides will be reviewed by Dr. Fitzhugh.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing orthopedic surgery for musculoskeletal tumors

Exclusion Criteria:

* pts who are pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing orthopedic surgery for remival of musculoskeletal tumors under general anesthesia
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
presence of tumor cells in the operative field | intraoperatively
  specimens taken twice from operative field; once just prior to removal of tumor and the second just after tumor removal.

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Gubenko, MD, Principal Investigator — UMDNJ/NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No